CLINICAL TRIAL: NCT04310254
Title: The Clinical Comparative Evaluation of Different Final Irrigation Protocols on Postoperative Endodontic Pain In Devital Teeth: A Prospective Randomized Clinical Trial
Brief Title: Effect of Different Final Irrigation Protocols on Postoperative Endodontic Pain in Devital Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 929
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Postoperative Pain; Endodontically Treated Teeth
Keywords: Endodontics; Postoperative Pain; Visual Analogue Pain Scale
MeSH Terms: conditions — Pain, Postoperative; Tooth, Nonvital | interventions — Edetic Acid

STUDY DESIGN:
Intervention Model Description: Parallel Assignment The patients were assigned to 3 medication groups randomly with an equal allocation rate between groups.The patients in the groups had same characteristics.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant and Outcomes Assessor) The patients were unaware as to which study group they had been allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EDTA and CHX solution (Active Comparator): Root canal irrigation was performed according to the guidelines to the manufacturers instructions for EDTA and CHX solution.
  Interventions: Procedure: EDTA and CHX Solution
- EDTA solution (Active Comparator): Root canal irrigation was performed according to the guidelines to the manufacturers instructions for EDTA solution.
  Interventions: Procedure: EDTA Solution
- CHX solution (Active Comparator): Root canal irrigation was performed according to the guidelines to the manufacturers instructions for CHX solution.
  Interventions: Procedure: CHX Solution

INTERVENTIONS:
Procedure: EDTA and CHX Solution — The teeth in this group were treated according to the guidelines for root canal treatment in single-session. The filling was removed and cavity was opened. After standart irrigation protocol, root canals were irrigated with Qmix 2in1 solution and obturated with gutta percha. Coronal restoration was complete using composite and/or fully crown if necessary.
  Arms: EDTA and CHX solution
Procedure: EDTA Solution — The teeth in this group were treated according to the guidelines for root canal treatment in single-session. The filling was removed and cavity was opened. After standart irrigation protocol, root canals were irrigated with EDTA solution and obturated with gutta percha. Coronal restoration was complete using composite and/or fully crown if necessary.
  Arms: EDTA solution
Procedure: CHX Solution — The teeth in this group were treated according to the guidelines for root canal treatment in single-session. The filling was removed and cavity was opened. After standart irrigation protocol, root canals were irrigated with CHX solution and obturated with gutta percha. Coronal restoration was complete using composite and/or fully crown if necessary.
  Arms: CHX solution

SUMMARY:
The purpose of this randomized clinical trial was to evaluate the incidence of postoperative pain after root canal treatment using different final irrigation protocols. Patients whom need root canal treatment for first time were included. The presence of postoperative pain was assessed after root canal treatment cases at 12, 24, 48, 72 hrs and 1 week.

DETAILED DESCRIPTION:
The aim of this clinical study was to evaluate the intensity and duration of postoperative pain following different final irrigation procedures. Patients who have asymptomaticdevital teeth required endodontic treatment were included in this study and routine root canal treatment procedure was applied to these teeth. All of the patients have been recruited from the Istanbul Medipol University Dental Clinics in Istanbul. Ninety asymptomatic teeth were randomly participated into 3 treatment groups in terms of intracanal medicament applied. The presence of postoperative pain was assessed after 12, 24, 48, 72 hrs and 1 week. Postoperative pain was recorded by each patient by using visual analogue pain scale. Before the treatments, the nature of the study, complications and associated risks were totally explained and written informed consent was obtained from all study participants. The patients were offered local anesthetic before the treatment start. The routine root canal treatment procedure was applied. Different final irrigation solutions applied in accordance to the manufacturers' instructions. At the end of treatment, each patient was given an evaluation sheet, explained the treatment procedure and using of visual analogue pain scales, and informed to be returned during the following one week. After one week the teeth was examined according to for pain intensity, percussion & palpation sensitivity, swelling, analgesic intake and clinical status.

ELIGIBILITY:
Inclusion Criteria:

-Patients who were healthy volunteers and who have devital premolar and molar teeth with PAI 3-5score requiring root canal treatment for first time.

Patients who were not included the study who;

* were pregnant or breast feeding during the duration of the study,
* have systemic disease, have any pain and/or any facial swelling, abscess,
* were immunocompromised,
* were under 18 yrs. and over 65 yrs. age,
* were taking antibiotics or corticosteroids within previous three days,
* have multiple teeth that required root canal treatment at the same time period; for eliminating pain referral,
* have root canals that could not be well-treated with orthograde root canal treatment.

Exclusion Criteria:

-The patients who forgot to fill out the form and took antibiotics and/or analgesics right after the first appointment of the therapy were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Postoperative Pain after Root Cana Treatment at 1 week. | Baseline, 12, 24, 48, 72 hours and 1 week.
  The primary outcome measure of the study was to assess if different intracanal medicaments and single-visit root canal treatment influence the occurrence of postoperative pain.Postoperative pain was assessed using a well defined Heft-Parker visual analogue scale (VAS) scale. Each patient recorded the pain level on a 100-mm VAS scale experimental basis for revising the graphic rating scale for pain in well-defined categories at 5 time intervals as 12, 24, 48, 72 hours and 1 week after treatment. The VAS scale was divided into 4 categories: No pain or faint pain corresponded to 0 mm. Mild pain was defined as greater than 0 mm and less than or equal to 25 mm. Mild pain included the descriptors of weak and mild pain. Moderate pain was defined as greater than 50 mm and less than 75 mm. Intense pain was defined as equal to or greater than 75 mm. Intense pain included the descriptors of strong, severe, and maximum possible.

CONTACTS AND LOCATIONS:
Overall Officials: Keziban Olcay, DDS, Phd, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)